CLINICAL TRIAL: NCT04189237
Title: Electroacupuncture Improves Pain and Wrist Functionality in Patients Undergoing Rehabilitation Therapy After Distal Radius Fracture
Brief Title: Electroacupuncture Improves Wrist Functionality and Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH108-REC1-141
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Electroacupuncture
Keywords: electroacupuncture; wrist functionality; distal radius fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture (Experimental): At the 4th week after surgery, electroacupuncture was performed, and the activity of wrist joint on the affected side was performed at same time, and at a frequency of two times per week for six weeks, for a total of twelve times.
  Acupoint selection: needles were inserted to Taixi (KI3), Taichong (LR3), Zusanli(ST36), Yanglingquan (GB34), contralateral to the operated leg and deqi sensation elicited at acupoints.
  Interventions: Other: Electroacupuncture
- Control group (No Intervention): At the 4th week after surgery, only the activity of wrist joint on the affected side was performed, and at a frequency of two times per week for six weeks, for a total of twelve times.

INTERVENTIONS:
Other: Electroacupuncture — needles were inserted to Taixi (KI3), Taichong (LR3), Zusanli(ST36), Yanglingquan (GB34), contralateral to the operated leg and deqi sensation elicited at acupoints.
  Arms: electroacupuncture

SUMMARY:
Electroacupuncture improves pain and wrist functionality in patients undergoing rehabilitation therapy after distal radius fracture Distal radius fracture is extremely common, and it is about 10% of all fractures in the human body. Therefore, the distal radius is the most frequently fractured part of the upper limbs of the human body. Once the fracture occurs, internal fixation is the main surgical procedure. And, the postoperative goal is to restore the function of the forearm and the mobility of the wrist joint. Therefore, rehabilitation treatment is the key. However, postoperative patients often delay rehabilitation therapy due to pain, resulting in stiffer wrist joints. In recent years, electroacupuncture(EA) has been widely used to relieve pain after surgery, and many studies have confirmed that it is effective. And it is already an alternative to postoperative pain relief. The investigators hope that by electroacupuncture, the investigators can help patients reduce pain, increase joint mobility, and make patients willing to start rehabilitation therapy, reduce joint stiffness, and restore wrist function as soon as possible, which will help patients return to work and normal life early.

Methods:

It is expected that 30 patients will be randomly assigned to the following groups: electroacupuncture group, control group without EA. Two groups of subjects started to rehabilitation at the 4th week after surgery.

DETAILED DESCRIPTION:
Electroacupuncture improves pain and wrist functionality in patients undergoing rehabilitation therapy after distal radius fracture Distal radius fracture is extremely common, and it is about 10% of all fractures in the human body. Therefore, the distal radius is the most frequently fractured part of the upper limbs of the human body. Once the fracture occurs, internal fixation is the main surgical procedure. And, the postoperative goal is to restore the function of the forearm and the mobility of the wrist joint. Therefore, rehabilitation treatment is the key. However, postoperative patients often delay rehabilitation therapy due to pain, resulting in stiffer wrist joints. In recent years, electroacupuncture(EA) has been widely used to relieve pain after surgery, and many studies have confirmed that it is effective. And it is already an alternative to postoperative pain relief. The investigators hope that by electroacupuncture, the investigators can help patients reduce pain, increase joint mobility, and make patients willing to start rehabilitation therapy, reduce joint stiffness, and restore wrist function as soon as possible, which will help patients return to work and normal life early.

Methods:

It is expected that 30 patients will be randomly assigned to the following groups: electroacupuncture group, control group without EA. Two groups of subjects started to rehabilitation at the 4th week after surgery.

Mode of operation: Electroacupuncture group: At the 4th week after surgery, electroacupuncture was performed, and the activity of wrist joint on the affected side was performed at same time, and at a frequency of two times per week for six weeks, for a total of twelve times.

Control group: At the 4th week after surgery, only the activity of wrist joint on the affected side was performed, and at a frequency of two times per week for six weeks, for a total of twelve times.

Acupoint selection: needles were inserted to Taixi (KI3), Taichong (LR3), Zusanli(ST36), Yanglingquan (GB34), contralateral to the operated leg and deqi sensation elicited at acupoints.

Data collection:

The evaluator does not know the patient group to achieve a single blind effect.

1. Use the visual analog scale (VAS) to assess the patient's pain level
2. Use the Disabilities of the Arm, Shoulder and Hand questionnaire(DASH) to assess the patient's pain and the functionality.
3. The degrees of wrist mobility were measured.
4. Three time points were recorded: before the first electroacupuncture (4th week after surgery, when removing fixation), after the 6th, 12th (last) electroacupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of distal radius fracture
* After internal fixation
* Age between 20 and 70 years old

Exclusion Criteria:

* serious heart rhythm
* epilepsy
* Severe pulmonary heart disease
* History of mental illness
* received acupuncture treatment 1 month ago

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-11-28 (Estimated); Study Completion 2020-11-28 (Estimated)

PRIMARY OUTCOMES:
Range of wrist motion | 4 weeks
  The degrees of wrist mobility measured with a goniometer, including flexion, extension, supination, pronation, ulnar deviation, radial deviation, and higher degrees mean a better outcome.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand(DASH) | 4 weeks
  Assess the patient's pain and the inability, the DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Cheng Chiu, MD, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, No. 2, Yude Rd, North District, Taichung City, Taiwan

IPD SHARING:
Plan to Share IPD: No